CLINICAL TRIAL: NCT00029393
Title: Induction of Stable Chimerism for Sickle Cell Anemia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Masking: None | Purpose: Treatment
Other Study IDs: 142; U01HL068091 (NIH)
Record Dates: First submitted 2002-01-10; First posted 2002-01-11 (Estimated); Last update posted 2016-07-29 (Estimated); Status verified 2008-01

CONDITIONS: Blood Disease; Hematopoietic Stem Cell Transplantation; Anemia, Sickle Cell
MeSH Terms: conditions — Hematologic Diseases; Anemia, Sickle Cell | interventions — Hematopoietic Stem Cell Transplantation; Immunosuppression Therapy

INTERVENTIONS:
Procedure: Hematopoietic Stem Cell Transplantation
Drug: Immunosuppression

SUMMARY:
To investigate a modified hematopoeitic cell transplantation (HCT) procedure for sickle cell disease that significantly reduces the toxicity of HCT, yet retains its therapeutic benefit.

DETAILED DESCRIPTION:
BACKGROUND:

Hematopoietic cell transplantation (HCT) has curative potential for individuals with sickle cell disease. While the results of conventional HCT have been good, this treatment carries risks of significant short- term and longterm toxicities. For this reason, HCT has been reserved for children who have experienced severe symptoms that predict a poor outcome. Of interest, some patients developed stable donor-host hematopoietic chimerism after conventional HCT. Due to a natural enrichment of donor erythrocytes in the blood, those who developed stable chimerism had a significant clinical benefit, even when there was a minority of donor cells. These observations have paralleled efforts to develop less-toxic, non-myeloablative preparative regiments for transplantation, proved first in a canine model of transplantation, and subsequently translated successfully in a clinical trial for older adults with hematological malignancies.

DESIGN NARRATIVE:

Multicenter open-label phase I-II study in 30 children with sickle cell disease that combines a non-myeloablative pre-transplant hematopoietic cell transplantation (HCT) therapy with modulated post-grafting immunosuppression to control host-versus-graft and graft-versus-host reactions. The approach relies on the ability to establish and maintain donor-host chimerism. The primary study endpoint is stable donor cell engraftment; secondary endpoints measure the impact of therapy on sickle cell-related symptoms and end-organ damage (disease-free survival, patient survival, graft-versus-host disease, complications etc). The trial will be conducted within the existing network of Comprehensive Sickle Cell Centers, and will be centrally coordinated by the Sickle Cell Coordinating Center.

ELIGIBILITY:
No eligibility criteria

Max Age: 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 2001-08; Primary Completion 2007-07 (Actual); Study Completion 2007-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mark Walters — UCSF Benioff Children's Hospital Oakland

REFERENCES:
- [Background] Walters MC, Patience M, Leisenring W, Rogers ZR, Aquino VM, Buchanan GR, Roberts IA, Yeager AM, Hsu L, Adamkiewicz T, Kurtzberg J, Vichinsky E, Storer B, Storb R, Sullivan KM; Multicenter Investigation of Bone Marrow Transplantation for Sickle Cell Disease. Stable mixed hematopoietic chimerism after bone marrow transplantation for sickle cell anemia. Biol Blood Marrow Transplant. 2001;7(12):665-73. doi: 10.1053/bbmt.2001.v7.pm11787529.
- [Background] Atkins RC, Walters MC. Haematopoietic cell transplantation in the treatment of sickle cell disease. Expert Opin Biol Ther. 2003 Dec;3(8):1215-24. doi: 10.1517/14712598.3.8.1215. PMID 14640947
- [Background] Iannone R, Casella JF, Fuchs EJ, Chen AR, Jones RJ, Woolfrey A, Amylon M, Sullivan KM, Storb RF, Walters MC. Results of minimally toxic nonmyeloablative transplantation in patients with sickle cell anemia and beta-thalassemia. Biol Blood Marrow Transplant. 2003 Aug;9(8):519-28. doi: 10.1016/s1083-8791(03)00192-7. PMID 12931121
- [Background] Horan JT, Liesveld JL, Fenton P, Blumberg N, Walters MC. Hematopoietic stem cell transplantation for multiply transfused patients with sickle cell disease and thalassemia after low-dose total body irradiation, fludarabine, and rabbit anti-thymocyte globulin. Bone Marrow Transplant. 2005 Jan;35(2):171-7. doi: 10.1038/sj.bmt.1704745. PMID 15531901